CLINICAL TRIAL: NCT02026583
Title: A Single Arm, Phase II Study of Simvastatin Plus XELOX and Bevacizumab as First-line Chemotherapy in Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor of Medicine, Sungkyunkwan University School of Medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB no : 2013-07-088
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Simvastatin

ARMS (1):
- Simvastatin (Experimental)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
1. Study Objectives 1) Primary Objective: Progression-free survival 2) Secondary Objectives:

   1. overall survival
   2. response rate
   3. incidence, nature and severity of all adverse events
   4. lipid lowering effect of simvastatin
   5. exploratory biomarker analysis : angiopoietin 2, BiP (Binding protein), Hsp (Heat shck protein) 90α
2. Study hypothesis In our recent in vitro study, addition of simvastatin to bevacizumab reduced proliferation, migration, invasion and tumor formation of endothelial cell. Moreover, colorectal cancer cell media which was treated with simvastatin combined with bevacizumab inhibited endothelial cell invasion and it was associated with decreased mediator of angiogenesis, such as angiopoietin 2, BiP and HSP 90α.. Treatment with bevacizumab and simvastatin more reduced the growth of xenograft tumors compared with bevacizumab alone.
3. Assessments 1) Safety : physical examination, vital signs, body weight, ECOG (Eastern Cooperative Oncology Group) performance status, clinical laboratory evaluation (chemistry, blood cell count) and any AE (adverse effect) graded by using CTCAE (Common Toxicity Criteria for Adverse Effects ) v 4.0 2) Efficacy : progression-free survival and overall survival will be collected. Response rate according to RECIST (Response Evaluation Criteria in Solid Tumors) 1,1 guideline will also be evaluated 3) PFS (Progression free survival): time from randomization to tumor progression or death 4) OS (Overall survival) : time from randomization to death or last follow-up 5) Biomarker analysis; The correlation between blood level, protein expression of angiopoietin 2, BiP, Hsp90α and clinical response will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed colorectal carcinoma
2. Stage IV or recurrent colorectal cancer
3. age ≥ 20 years
4. ECOG performance status ≤1
5. At least one measurable tumor mass according to RECIST 1.1
6. Expected survival for approximately 12 weeks or longer
7. No prior systemic chemotherapy
8. At least 4 weeks later after surgery or radiotherapy
9. At least 12 months after adjuvant chemotherapy

Exclusion Criteria:

1. Prior statins therapy within 1-year from the date of study entry
2. Prior chemotherapeutic treatment for metastatic colorectal cancer.
3. Prior other anti-VEGF (vascular endothelial growth factor) or TKIs (Tyrosine kinase inhibitors) treatment
4. Current, Known CNS(central nervous system) malignancy (history of completely resected or irradiated brain metastases by WBRT (whole-brain radiation therapy) or stereotactic radiosurgery allowed.
5. Severe or unstable cardiac disease, including (for example) coronary artery disease requiring increased doses of anti-anginal medication and/or coronary angioplasty (including stent placement) within the preceding 24 months(congestive heart failure NYHA (New York Heart Association) III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)
6. Past or current history (within the last 5 years prior to treatment start) of other malignancies except metastatic colorectal cancer (Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible)
7. Uncontrolled systemic illness such as DM (diabetes mellitus), hypertension, hypothyroidism and infection
8. History of thromboembolic or hemorrhagic events within 6 months prior to treatment
9. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to enrollment.
10. Evidence of bleeding diathesis or coagulopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Progression free survival | During treatment : up to 6weeks, off the treatment : up to 8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea